CLINICAL TRIAL: NCT02133248
Title: Identification of Donor Specific B Cells Will Positively Affect Monitoring and Treatment of Donor Specific Antibodies and Antibody Mediated Rejection
Brief Title: Identification of Donor Specific B Cells and Antibody Mediated Rejection
Status: Terminated | Type: Observational
Why Stopped: enrollment issues due to COVID-19 related research suspension and PI left the institution
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0076; A534280 (Other: UW Madison); SMPH\MEDICINE\NEPHROLOGY (Other: UW Madison)
Record Dates: First submitted 2014-05-05; First posted 2014-05-08 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Sensitized Kidney Transplant Recipients
Keywords: donor specific antibodies; B cells; antibody mediated rejection; kidney transplant; desensitization

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen peripheral blood mononucleated cells and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- kidney recipient waitlist: Subjects on waitlist for Kidney transplant who are sensitized
- chronic antibody mediated rejection: Kidney transplant recipient who are diagnosed with chronic antibody mediated rejection
- control: Normal subjects-no kidney transplant or chronic rejection

SUMMARY:
Many people who are on the wait list for a kidney transplant have harmful antibodies, called donor specific antibodies (DSA), which will attack foreign tissue such as the transplanted organ. These people are considered to be"sensitized". Prior to receiving a kidney, these patients undergo desensitization treatments to remove these harmful antibodies. Levels of DSA are measured after desensitization, but the cells that produce the DSA, donor specific B cells (DSB), have not generally been measured. Additionally, if a person experiences chronic rejection due to antibodies they are also desensitized, but only the DSA are measured. This study will measure the DSA and, using new techniques, the DSB in two study groups: those who are receiving an organ and those experiencing chronic antibody mediated rejection after receiving an organ. The hypothesis is people with higher levels of DSB after desensitization are more likely to develop antibody mediated rejection.

DETAILED DESCRIPTION:
Patients that are sensitized, who have panel reactive antibodies (PRAs) > 20%, comprise a disproportionate and increasing cluster on the wait list (33%), and have to wait longer to receive a transplant than non-sensitized patients. By 36 months on the wait list, 10% died before receiving a transplant. Those who do receive transplants require desensitization. The current desensitization protocols include anti-CD20 monoclonal antibody to remove B cells, a proteasome inhibitor to eliminate plasma cells and plasma exchange and/or intravenous immunoglobulin (IVIG) to remove pre-formed donor specific antibodies (DSA). The success of these protocols can be measured using single antigen bead (SAB) luminex technology. These desensitization protocols have been shown to significantly decrease mean fluorescence intensity (MFI). Desensitization protocols typically are more effective in removing antibodies that recognize HLA Class I molecules than those that recognize HLA Class II molecules. Unfortunately, even after pre-conditioning, sensitized patients are more likely to develop antibody mediated rejection (ABMR) than patients that do not have donor specific antibodies prior to transplant. Currently, serum levels of DSA are measured after desensitization, but not donor specific B cells (DSB). It is possible that B cells and/or plasma cells remain after treatment. Donor specific B cells, upon transplant and the accompanying exposure to antigen, can be re-stimulated to both produce antibody and also to develop into plasma cells which produce antibody. Therefore, potentially a better means of determining whether desensitization has been successful would be to look at both the DSA level using SAB technology as described above and to look at DSB to determine if these cells have been adequately cleared by the desensitization protocol.

Specific Aim 1 Hypothesis: Patients who have adequate clearance of serum DSA, but who still have significant populations of DSB are more likely to develop ABMR.

In Specific Aim 1, the investigators will utilize cutting edge technology to observe levels of anti-HLA antibodies, particularly donor specific antibodies, present in sensitized patients by staining DSB with HLA class I tetramers. This method allows enumeration and characterization of the source of DSA, the DSB. The investigators will determine the number of DSB and donor specific plasma cells (DSPC) prior to and after desensitization as well as later post transplant. In addition, the investigators will look at the phenotype and activation state of the DSB prior to transplant and after transplant. HLA class I tetramers are MHC class I molecules of a particular allele which are refolded with a peptide in the peptide binding groove, biotinylated on the C terminal tail and tetramerized using streptavidin conjugated to a fluorophore such as phycoerythrin (PE). Similarly, HLA class II tetramers are made of MHC class II alleles. B cells retain membrane bound antibody which has the exact specificity of the soluble antibodies that it also produces. The tetramers will bind only to B cells that have antibodies against that specific HLA class I allele on the surface, since the binding is determined only by the specificity of the antibody. At the same time, the cells will be stained with other markers to determine the activation state and phenotype of the DSB. This assay is done using flow cytometry. Additionally, the investigators will measure BAFF and APRIL cytokine levels by Elisa at all time points. These cytokines are closely related to B cell development. There is data to suggest that BAFF is elevated after some forms of desensitization, which could enhance new B cell development.

Specific Aim 1 Hypothesis: Patients who have adequate clearance of serum DSA, but who still have significant populations of DSB are more likely to develop ABMR.

In Specific Aim 1, the investigators will utilize cutting edge technology to observe levels of anti-HLA antibodies, particularly donor specific antibodies, present in sensitized patients by staining DSB with HLA class I tetramers. This method allows enumeration and characterization of the source of DSA, the DSB. The investigators will determine the number of DSB and donor specific plasma cells (DSPC) prior to and after desensitization as well as later post transplant. In addition, the investigators will look at the phenotype and activation state of the DSB prior to transplant and after transplant. HLA class I tetramers are MHC class I molecules of a particular allele which are refolded with a peptide in the peptide binding groove, biotinylated on the C terminal tail and tetramerized using streptavidin conjugated to a fluorophore such as phycoerythrin (PE). Similarly, HLA class II tetramers are made of MHC class II alleles. B cells retain membrane bound antibody which has the exact specificity of the soluble antibodies that it also produces. The tetramers will bind only to B cells that have antibodies against that specific HLA class I allele on the surface, since the binding is determined only by the specificity of the antibody. At the same time, the cells will be stained with other markers to determine the activation state and phenotype of the DSB. This assay is done using flow cytometry. Additionally, we will measure BAFF and APRIL cytokine levels by Elisa at all time points. These cytokines are closely related to B cell development. There is data to suggest that BAFF is elevated after some forms of desensitization, which could enhance new B cell development.

The investigators will obtain a blood draw from subjects once consent is obtained and utilize this sample to establish a baseline of B cells that produce antibodies that recognize HLA class I tetramers of the same type as those previously identified by SAS anti-HLA antibody analysis. Immediately prior to and after the patient receives a transplant, the SAB anti-HLA antibody analysis, tetramer analysis, and BAFF/APRIL Elisas will be repeated. Analyses will also be performed between 6 weeks and 2 months after transplant.

Specific Aim 2 Hypothesis: During chronic rejection, patients who respond well to desensitization and who are able to maintain tolerance after desensitization will have fewer residual DSB.

In Specific Aim 2, the investigators will utilize the same technology to quantify and characterize DSA and DSB when a patient experiences chronic rejection due to ABMR. In this case, the patient may not have had DSA when transplanted, but developed de novo DSA (dnDSA) after transplant, causing rejection. Or the patient may have had DSA, been desensitized successfully, maintained tolerance for a period of time, then either lost tolerance or developed dnDSA. The timelines will be similar to specific aim 1 - the investigators will take samples at the following timepoints: upon diagnosis of ABMR, 1 week after desensitization, then 2 to 3 months after desensitization to look for rebound.

In addition to enrollment of new subjects, the investigators will also enroll healthy normal individuals to serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 inclusive
* Patients on UWHC Kidney Transplant waitlist identified as sensitized or
* UWHC kidney transplant recipient patients diagnosed with antibody mediated rejection

Exclusion Criteria:

* Inability to provide informed consent to participate in study
* Diagnosed with an autoimmune disorder or kidney problems, currently on immunosuppressive or immunomodulatory medication, or any current malignancies (healthy controls only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aim 1: Subjects on the wait list for kidney transplantation who are patients of the University of Wisconsin Hospital and Clinics (UWHC) and are identified as sensitized Aim 2: Kidney transplant recipients who are having a clinically indicated biopsy due to suspected antibody mediated rejection and are patients of the UWHC Both aims: Control subjects recruited from the University of Wisconsin Office of Clinical Trials control recruitment database
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Donor specific B (DSB) cell populations are reduced after desensitization. | 1 week post desensitization treatment
  The primary objective of this study is to determine whether desensitization results in not only a decrease in anti-HLA antibodies, but also a decrease in donor specific B cell populations.
Donor specific B (DSB) cell populations are reduced after desensitization. | 6 weeks-3 months post desensitization
  The primary objective of this study is to determine whether desensitization results in not only a decrease in anti-HLA antibodies, but also a decrease in donor specific B cell populations.

SECONDARY OUTCOMES:
Correlation of DSB to incidence of antibody mediated rejection | 12 months post desensitization
  The secondary objective of this study is to correlate numbers and/or phenotypes of DSB remaining after desensitization to occurrence, for transplant recipients) or recurrence (for recipients with chronic antibody mediated rejection (ABMR)) of ABMR.
B-cell activating factor (BAFF) levels increase after desensitization | 1 week post desensitization
  Determine whether BAFF levels are increased in sensitized subjects, as well as to determine if this cytokines are increased post desensitization, as has been suggested in the literature.
B-cell activating factor (BAFF) levels increase after desensitization | 6 weeks-3 months post desensitization
  Determine whether BAFF levels are increased in sensitized subjects, as well as to determine if this cytokines are increased post desensitization, as has been suggested in the literature.
A proliferation inducing ligand (APRIL) levels increase after desensitization | 1 week post desensitization
  Determine whether APRIL levels are increased in sensitized subjects, as well as to determine if this cytokines are increased post desensitization, as has been suggested in the literature.
A proliferation inducing ligand (APRIL) levels increase after desensitization | 6 weeks-3 months post desensitization
  Determine whether APRILlevels are increased in sensitized subjects, as well as to determine if this cytokines are increased post desensitization, as has been suggested in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Arjang Djamali, MD, Principal Investigator — University of Wisconsin Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Niederhaus SV, Muth B, Lorentzen DF, Wai P, Pirsch JD, Samaniego-Picota M, Leverson GE, D'alessandro AM, Sollinger HW, Djamali A. Luminex-based desensitization protocols: the University of Wisconsin initial experience. Transplantation. 2011 Jul 15;92(1):12-7. doi: 10.1097/TP.0b013e31821c93bb. PMID 21512428
- [Background] Lobashevsky AL, Higgins NG, Rosner KM, Mujtaba MA, Goggins WC, Taber TE. Analysis of anti-HLA antibodies in sensitized kidney transplant candidates subjected to desensitization with intravenous immunoglobulin and rituximab. Transplantation. 2013 Jul 27;96(2):182-90. doi: 10.1097/TP.0b013e3182962c84. PMID 23778648
- [Background] Djamali A, Muth BL, Ellis TM, Mohamed M, Fernandez LA, Miller KM, Bellingham JM, Odorico JS, Mezrich JD, Pirsch JD, D'Alessandro TM, Vidyasagar V, Hofmann RM, Torrealba JR, Kaufman DB, Foley DP. Increased C4d in post-reperfusion biopsies and increased donor specific antibodies at one-week post transplant are risk factors for acute rejection in mild to moderately sensitized kidney transplant recipients. Kidney Int. 2013 Jun;83(6):1185-92. doi: 10.1038/ki.2013.44. Epub 2013 Feb 27. PMID 23447068
- [Background] Tait BD, Susal C, Gebel HM, Nickerson PW, Zachary AA, Claas FH, Reed EF, Bray RA, Campbell P, Chapman JR, Coates PT, Colvin RB, Cozzi E, Doxiadis II, Fuggle SV, Gill J, Glotz D, Lachmann N, Mohanakumar T, Suciu-Foca N, Sumitran-Holgersson S, Tanabe K, Taylor CJ, Tyan DB, Webster A, Zeevi A, Opelz G. Consensus guidelines on the testing and clinical management issues associated with HLA and non-HLA antibodies in transplantation. Transplantation. 2013 Jan 15;95(1):19-47. doi: 10.1097/TP.0b013e31827a19cc. PMID 23238534